CLINICAL TRIAL: NCT02926963
Title: Generation of Powerful Biological Tools - Fibroblast or Inducible Pluripotent Bone Marrow Cells - for Understanding the Pathophysiology of Chronic Granulomatous Disease.
Brief Title: Generation of Powerful Biological Tools for Understanding the Pathophysiology of Chronic Granulomatous Disease.
Acronym: FIBRO CGD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 38RC09.018; 2009-A00944-53 (Other: ID RCB)
Record Dates: First submitted 2016-10-04; First posted 2016-10-06 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Chronic Granulomatous Disease
Keywords: Chronic Granulomatous Disease, Nox2, p22phox, iPS cells
MeSH Terms: conditions — Granulomatous Disease, Chronic; Granulomatous Disease, Chronic, Autosomal Recessive, Cytochrome B-Negative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chronic Granulomatous Disease (Experimental): Sample collection were performed from patients with chronic granulomatous disease linked to X or due to Autosomal Recessive (AR) forms AR220, AR470 and AR670.
  Interventions: Other: samples collection : hair and skin biopsy

INTERVENTIONS:
Other: samples collection : hair and skin biopsy

SUMMARY:
Chronic granulomatous disease (CGD) is a rare genetic disease of innate immune due to the malfunction of phagocytic cells unable to destroy pathogens during infection. The four genes implicated are CYBB, CYBA, NCFA and NCF2 respectively encoding Nox2, p22phox, p47phox and p67phox. Nox2 analogs have recently been discovered in cells other than phagocytes. So the question arises on physiopathological impact of the absence of theses proteins not only in phagocytes but also in other cells types such as fibroblasts or neurons.

The principal objective is thus to study the impact of protein deficits Nox2 and p22phox, in the pathophysiology of neurons from inducible pluripotent bone marrow cells (iPSC).

For this purpose, a collection was built of fibroblasts and keratinocytes from patients with different forms of CGD to get iPSC similar to embryonic marrow cells and differentiable into several cell types (neurons, phagocytes).

DETAILED DESCRIPTION:
Non randomised pilot descriptive multicentric study. Since recently it has been shown that Nox2p22phox protein is expressed not only in phagocytic cells but also in non-phagocytic cells such as fibroblasts, epithelial cells ,vascular cells, neurons. If pathological consequences of the deficiency Nox2 and p22phox, essential to the production of bactericidal toxic derivatives at the level of phagocytic cells, is well documented, impact of their absence in other types of non-phagocytic cells is not known. A better understanding of the impact of the absence of these proteins in these tissues could improve the management of CGD patients by providing a more specific monitoring of their condition. Similarly the formation of different cell models of all genetic forms of CGD that do not exist at present will be of great use to study the physiopathology of this disease and as tools for future studies.

The study requires the inclusion of minor subjects as CGD is usually diagnosed in early childhood ( <2 years), it is rare (frequency 1/200 000) and the life expectancy is reduced.

To elaborate the cells collection, hair and skin biopsy are necessary. They will be performed under local anesthesia for adults, and during a planned general anesthesia for minors.

Fibroblasts and keratinocytes in culture will be obtained by conventional control methods and the absence of expression of p22phox or Nox2 will be checked.

Measurement of the kinetics of neuronal development and apoptosis iPSC will be performed in a differentiation system 2 dimensions on stromal cells MS5. For that, markers of neuronal differentiation of each step will be measured.

Measurement of Reactive Oxygen Species (ROS) in phagocytes and p22phox deficient Nox2 from differentiation from iPSC (chemiluminescence, flow cytometry) will be performed.

Measurement of the effectiveness of phagocytosis (phagocytic function) in phagocytes deficient p22phox and Nox2 from differentiation from iPSC (flow cytometry) will be performed.

The absence of protein and p22phox Nox2 in phagocytes and p22phox deficient Nox2 from differentiation from the iPSC (western blot, flow cytometry) will be verified.

Kinetic of transformation of fibroblasts derived from CGD patients with deficiency or p22phox Nox2 in myofibroblasts will be measured.

To answer the principal objective of this study the recruitment of 10 patients will be necessary.

ELIGIBILITY:
Inclusion Criteria:

* diagnostic of chronic granulomatous disease (CGD) with determined genetic form
* for minors, patient requiring installation or removal of deep venous general anesthesia.

Exclusion Criteria:

* patients with acute infections scalable to practice of skin biopsy under local anesthesia
* patient with impaired hemostasis acquired (drug) or innate.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-10; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
to study the impact of protein deficits Nox2 and p22phox, in the physiopathology of neurons from inducible pluripotent bone marrow cells (iPSC) | one year
  measurement of the kinetics of neuronal differentiation and identification of subtypes cell formed

SECONDARY OUTCOMES:
To study the impact of protein deficits Nox2 and p22phox on cytochrome b558 synthesis process of phagocytes from inducible pluripotent bone marrow cells ( iPSC ). | 6 months
  Evaluation of the synthesis of cytochrome b558 by phagocytes from the transformation of iPSC as a cellular model for studying the impact of the lack of p22phox and Nox2
To study the impact of protein deficits Nox2 and p22phox , at the physiology of fibroblasts and their transformation into myofibroblasts | two years
  Measuring markers of transformation of fibroblasts into myofibroblasts
Constitute cellular models of different types of CGD for future physiopathological studies and therapeutic trials | for years
  Get neutrophils and monocytes from the iPSC having the characteristics of human neutrophils of different genetic forms of CGD

CONTACTS AND LOCATIONS:
Overall Officials: Dominique PLANTAZ, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble Alpes, Grenoble, Cs10217, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Neill S, Brault J, Stasia MJ, Knaus UG. Genetic disorders coupled to ROS deficiency. Redox Biol. 2015 Dec;6:135-156. doi: 10.1016/j.redox.2015.07.009. Epub 2015 Jul 17. PMID 26210446
- [Background] Bedard K, Krause KH. The NOX family of ROS-generating NADPH oxidases: physiology and pathophysiology. Physiol Rev. 2007 Jan;87(1):245-313. doi: 10.1152/physrev.00044.2005. PMID 17237347
- [Background] Nakano Y, Longo-Guess CM, Bergstrom DE, Nauseef WM, Jones SM, Banfi B. Mutation of the Cyba gene encoding p22phox causes vestibular and immune defects in mice. J Clin Invest. 2008 Mar;118(3):1176-85. doi: 10.1172/JCI33835. PMID 18292807
- [Background] Schiavone S, Sorce S, Dubois-Dauphin M, Jaquet V, Colaianna M, Zotti M, Cuomo V, Trabace L, Krause KH. Involvement of NOX2 in the development of behavioral and pathologic alterations in isolated rats. Biol Psychiatry. 2009 Aug 15;66(4):384-92. doi: 10.1016/j.biopsych.2009.04.033. Epub 2009 Jun 26. PMID 19559404
- [Background] Brault J, Goutagny E, Telugu N, Shao K, Baquie M, Satre V, Coutton C, Grunwald D, Brion JP, Barlogis V, Stephan JL, Plantaz D, Hescheler J, Krause KH, Saric T, Stasia MJ. Optimized Generation of Functional Neutrophils and Macrophages from Patient-Specific Induced Pluripotent Stem Cells: Ex Vivo Models of X(0)-Linked, AR22(0)- and AR47(0)- Chronic Granulomatous Diseases. Biores Open Access. 2014 Dec 1;3(6):311-26. doi: 10.1089/biores.2014.0045. PMID 25469316